CLINICAL TRIAL: NCT01990365
Title: The Influence of Vertebral Mobility on Low Back Pain in Patients With Acute Osteoporotic Vertebral Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: TH No 6-3
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporotic Vertebral Fracture
Keywords: Vertebral fracture, low back pain, gips, mobility
MeSH Terms: conditions — Spinal Fractures; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many patients with acute osteoporotic vertebral fracture (acute OVFs) admitted because of low back pain. But there are only part of patients with acute OVFs, because some patients do not have low back pain although OVFs occurred.

DETAILED DESCRIPTION:
Many patients of acute OVFs present with low back pain. While there are also many patients without low back pain even if acute OVFs occurred. The mechanism of low back pain after acute OVFs is well unknown. We set up a hypothesis that low back pain results from vertebral body mobility, which refers to a change of vertebral height or configuration with changes in body positioning. The main objective of this study is to reveal the relationship between vertebral body mobility and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute osteoporosis fractures

Exclusion Criteria:

* Patients without acute osteoporosis fractures (metastasis, infection, deformity,etc)

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporotic patients with acute vertbral fracture
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Relationship between dynamic mobility of acute vertebral fracture body and low back pain | Up to 36 months
  The investigators plan to analyze 300 patients who presented with acute back pain and were diagnosed as having acute OVFs on MRI.
  All radiographs were taken at the initial visit. Fracture mobility was determined by comparing cross-table supine lateral radiographs with sitting lateral radiographs (dynamic radiography). Mobility was considered present when a measurable change in vertebral body height occurred between supine and sitting radiographs.We also evaluate low back pain using visual analog scale (VAS) score.
  Then the patients undergo external fixation using Gips. After Gips fixation, dynamic radiography was performed again to evaluate reduction of dynamic mobility of the OVF body. VAS score was also evaluated after external fixation.
  We investigate patients' background such as age, sex, bone mineral density, etc.
  We performed statical analyses to determine the factors which related to low back pain after acute OVFs, especially fracture mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan